CLINICAL TRIAL: NCT00736450
Title: Investigator Initiated Pilot Study of Microarray Directed Therapy for Diffuse Large B-cell Lymphoma Using Genasense With CHOP-R
Brief Title: Oblimersen Sodium & Combination Chemotherapy in Treating Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Manufacturer is no longer making the drug.
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0462-07-FB; NCI-2009-01692 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — oblimersen; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Biopsy; Microarray Analysis; Gene Expression Profiling; Immunohistochemistry; Cytogenetic Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Biological: oblimersen sodium; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Procedure: biopsy; Genetic: microarray analysis; Other: immunohistochemistry staining method; Genetic: gene expression analysis; Genetic: cytogenetic analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Procedure: biopsy — Correlative studies
  Other Names: biopsies
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: gene expression analysis — Correlative studies
Genetic: cytogenetic analysis — Correlative studies

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Oblimersen sodium may help chemotherapy work better by making cancer cells more sensitive to the drugs. Giving oblimersen sodium together with combination chemotherapy may kill more cancer cells. PURPOSE: This clinical trial is studying the side effects of giving oblimersen sodium together with combination chemotherapy and to see how well it works in treating patients with newly diagnosed stage I, stage II, stage III, or stage IV diffuse large B-cell lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To assess the feasibility and determine the rate of rapid turn around, that is within 7 working days of receipt of adequate tissue at UNMC for a AFFYmetrix microarray study of newly diagnosed patients with Diffuse Large B-cell Lymphoma (DLBCL) who will then receive treatment on this protocol. II. To evaluate efficacy (complete response rate) of Genasense (antisense bcl-2) given in addition to standard cyclophosphamide, vincristine, doxorubicin, and prednisone -rituximab (CHOP-R) to newly diagnosed patients with DLBCL who are found to have the ABC type after gene expression profiling or IHC as compared to newly diagnosed patients with DLBCL who do not express the ABC type that go on to receive standard CHOP-R (control). III. To evaluate the toxicity of Genasense (antisense bcl-2) given in addition to standard cyclophosphamide, vincristine, doxorubicin, and prednisone -rituximab (CHOP-R) for newly diagnosed patients with DLBCL who are found to have the ABC type after gene expression profiling. OUTLINE: Patients with diffuse large B-cell lymphoma (DLBCL) that expresses ABC type proceed to treatment in group I. Patients with DLBCL that does not express ABC type proceed to treatment in group II. GROUP I (oblimersen sodium and standard CHOP-R): Patients receive oblimersen sodium IV continuously on days 1-7. Patients also receive CHOP-R comprising rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 5 and prednisone orally on days 5-10. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. GROUP II (standard CHOP-R alone): Patients receive CHOP-R comprising rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1 and prednisone orally on days 1-5. Treatment repeats every 3 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with Diffuse Large B-cell Lymphoma (DLBCL) (any stage) OR composite lymphoma with >= 50% DLBCL
* Adequate diagnostic tissue for microarray gene expression analysis or IHC analysis
* Karnofsky Performance Status >= 70 (ECOG 0, 1)
* No prior chemotherapy (with the exception of 1 cycle CHOP-R based on current diagnosis, clinical condition, and availability/feasibility of initiating Genasense), immunotherapy, radiotherapy, or investigational therapies for NHL; steroid therapy is allowed only if required for maintenance of another chronic disease (e.g., rheumatoid arthritis)
* Patients aged >= 60 years, or patients with a history of coronary artery disease, congestive heart failure, hypertension, diabetes, or hyperlipidemia must have an estimated ejection fraction >= 0.45 (45%) by MUGA or echocardiography, performed within two months of study entry
* Patients must be willing to give written informed consent, and sign an institutionally approved consent form prior to initiating genasense or any study related activities (i.e., Genasense & microarray)
* Females of childbearing potential must have a negative serum pregnancy test prior to enrollment in the study
* Adequate venous access for 7-day continuous infusion
* Patients without evidence of severe organ dysfunction as determined within two weeks of 1st cycle of CHOP-R: 1) Hemoglobin > 8 g/dl; 2) Absolute neutrophil count > 1000/; 3) Platelets > 100,000 (lower blood counts may be acceptable if due to lymphoma after review with principal investigator); 4) Creatinine =< 2.0 mg/dL (unless due to NHL); 5) Bilirubin =< 2.0 mg/dL; 6) AST =< 3 x upper normal; 7) ALP =< 3 x upper normal (unless due to NHL)
* Men and women of reproductive potential must agree to use TWO of the following forms of birth control every time they have sex throughout the study and for up to 3 months following discontinuation of study drug: hormonal birth control methods, condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicidal, IUD, or surgical sterilization while participating in this study

Exclusion Criteria:

* Significant medical disease other than cancer including: 1) Any bleeding or coagulation disorder including a history of autoimmune hemolytic anemia or autoimmune thrombocytopenia; 2) Severe pulmonary disease; 3) Uncontrolled congestive heart failure; 4) New York Heart Association class III or IV disease; 5) Uncontrolled seizure disorder; and 6) Active infections
* Less than 3 weeks from prior major surgery
* Prior organ allograft
* Known HIV infection (due to expected frequent occurrence of myelo-suppression and immunosuppression)
* Women who are pregnant (confirmed by a serum pregnancy test in females of reproductive potential) or breast-feeding (women of child-bearing potential and sexually active males must be advised to take precautions to prevent pregnancy during treatment or remain abstinent)
* Women of child-bearing potential and sexually active males must be advised to take precautions to prevent pregnancy during treatment (unless the subject or subject's partner(s) is sterile, i.e., women who have had a hysterectomy or have been post-menopausal for at least twelve consecutive months) or remain abstinent
* Known hypersensitivity to phosphorothiate-containing oligonucleotides
* Concurrent investigational, corticosteroid therapy or any other anti-cancer treatments (such as chemotherapy, radiation, biologic or investigational therapies) while receiving protocol therapy; other than one cycle CHOP-R allowed based on current diagnosis, clinical condition, and availability/feasibility of initiating Genasense; other than chronic steroid use for another indication (For stage I/II or as clinically indicated- involved field irradiation as per standard practice is accepted)
* Other investigational drug therapy within 30 days of study entry
* Secondary leukemia or history of antecedent hematologic disorder
* History of second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for three or more years)
* No active CNS disease defined as symptomatic meningeal lymphoma or known CNS parenchymal lymphoma
* Concomitant anticoagulant therapy is not permitted (with the exception of 1 mg/day of warfarin for central line prophylaxis)
* Known hypersensitivity to G3139 (Genasense) or R-CHOP
* Neurologic disorders, overt psychosis, mental disability or evidence of limited capacity to provide fully informed consent or cooperation with the complexities of the treatment program

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-07-23 (Actual); Primary Completion 2012-10-09 (Actual); Study Completion 2012-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD MBA, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - Saint Francis Medical Center, Grand Island, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 37 subjects consented, 19 were Not ABC gene type positive so were removed from the study.
  Of the 18 remaining eligible, 4 patients opted for standard of care and withdrew from the study.
  13 subjects had microarray analysis conducted with tissue.
Groups:
- Arm I: Patients in this study who are found to have the Activated B-Cell (ABC) type after gene expression profiling or Immunohistochemistry (IHC) staining will receive combination chemotherapy with the standard CHOP-R with Genasense (oblimersen) (anti-bcl2 oligonucleotide).
  oblimersen sodium: Given IV
  rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate: Given IV
  prednisone: Given orally
Period: Overall Study
Arm/Group | Arm I
Started | 37
Completed | 12
Not Completed | 25
Not completed — Not ABC gene eligible | 19
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] — Population: The mean age was calculated from only the 14 subjects that received study treatment.
  years
    number analyzed (Participants) | 14
    (all) | 53 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Time to Perform Microarray Study After Receipt of Tissue
Description: The time from tissue harvest to release of microarray test and IHC assay results will be noted in days.
Time Frame: Upto 14 days
Measure: Mean (Full Range); unit: days
Arm/Group | Arm I
Number analyzed (Participants) | 13
days | 4.4 [0 to 14]

2. Primary Outcome: Number of Participants With Microarray Testing Results Are Completed Within 7 Days.
Time Frame: Upto 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 13
Participants
  results within 7 days or less | 11
  results in more than 7 days | 2

3. Secondary Outcome: Efficacy of Treatment, in Terms of Complete Response Rate (Anyone Achieving a CR or Cru)
Description: Response criteria are the recommendations of the International Harmonization Project's update to the International Working Group guidelines. Complete response (CR) is defined as disappearance of all evidence of disease; Partial response (PR) is defined as regression of measurable disease and no new sites
Time Frame: End of treatment, an average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 13
Participants
  complete response | 12
  partial response | 1

ADVERSE EVENTS:
Time Frame: Participants adverse event data was collected from time of initial study drug dosing until completed study treatment. (approximately 6 months)
Description: Only reporting all Serious adverse events and Other AEs grade 3 and 4.
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=14)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Platelet count decreased (Investigations) | 1 (3) — thrombocytopenia
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
confusion (Psychiatric disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cells decreased (Investigations) | 1 (2) — Leukocyte count decreased
Urinary tract infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=14)
White blood cell decreased (Investigations) | 10 (22) — leukocytes
Neutrophil count decreased (Investigations) | 10 (36)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) — Thrombus- right arm related to PIC line.
Infusion related reaction (General disorders) | 1 (1) — reaction to rituxan
Infections and infestations - Other (Infections and infestations) | 1 (1) — oral infection
Thromboembolic event (Vascular disorders) | 1 (1) — deep vein thrombosis
anemia (Blood and lymphatic system disorders) | 2 (2) — low hemoglobin
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased (Infections and infestations) | 4 (6)
Constipation (Gastrointestinal disorders) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) — infection, port site
Infections and infestations - Other (Infections and infestations) | 1 (1) — opportunistic infection
Headache (Nervous system disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) — maxillary
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
lymphocyte count decreased (Investigations) | 1 (5)
sepsis (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes